CLINICAL TRIAL: NCT01325259
Title: Molecular Imaging of Cerebral Amyloid Plaques Using PET With Fluoro Tracker for Early Diagnosis of Alzheimer's Disease
Brief Title: FluoroAv45 Imaging Research-in Alzheimer's Disease
Acronym: FAIR-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PHRN08-VC / FAIR AD
Record Dates: First submitted 2011-02-21; First posted 2011-03-29 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alzheimer's disease (Experimental): 30 patients suffering from Alzheimer's disease
  Interventions: Other: neuropsychologic assessment; Radiation: [18F]AV-45 PET; Radiation: 18-FDG PET; Other: MRI
- Mild Cognitive Impairment (Experimental): 20 patients suffering from Mild Cognitive Impairment
  Interventions: Other: neuropsychologic assessment; Radiation: [18F]AV-45 PET; Radiation: 18-FDG PET; Other: MRI
- Control (Experimental): 15 subjects with no cognitive impairment
  Interventions: Other: neuropsychologic assessment; Radiation: [18F]AV-45 PET; Radiation: 18-FDG PET; Other: MRI

INTERVENTIONS:
Other: neuropsychologic assessment — Mini Mental Status Examination, Mattis dementia rating scale, Geriatric Depression Scale, Edinburgh Inventory, DO 80, 12 irregular words dictation, RL-RI16, DMS 48, Rey complex figure, Stroop test, span right and reverse, praxis, ESR words, ESR drawings, Trail Making Test A and B, code test from WAIS III, Hayling inhibition test, fluences, NPI
Radiation: [18F]AV-45 PET — intravenous injection of 4 MBq/kg of [18F]AV-45
Radiation: 18-FDG PET — intravenous injection of 100 to 120 MBq of FDG
Other: MRI — Magnetic Resonance Imaging

SUMMARY:
Rationale: improving the early detection of AD at prodromal pre-dementia stages has become a major matter of concern. There is now an important body of literature stating that early isolated cognitive deficits (Mild Cognitive Impairment-MCI-) predict the risk of developing AD. Several biomarkers are now available : specific and sensitive neuropsychological assessments, morphometric evaluation of hippocampal volume and white matter changes by MRI, cerebrospinal fluid or plasma dosage of Ab fragments and tau proteins, assessment of brain glucose hypometabolism in temporo-parietal regions with PET [F18]FDG. However, PET imaging using labelled compounds specifically binding to APs has been suggested to improve the diagnostic reliability and to potentially help in shortening the delay until formal clinical diagnosis of AD. F18 AV45 is a new radiotracer which kinetics characteristics allows 10 to 15 minutes acquisition 50 to 60 minutes post injection.

Objectives: The primary objective of the study is to compare F18 AV45 cortical uptake in AD, MCI patients and Healthy Controls.

Secondary objectives will be to compare cortical uptake of F18 AV45 in MCI subject who will have convert toward dementia versus those who will not, at two year follow-up period, to compare level of 18F-AV45 cortical uptake with neuropsychological testing, PET FDG hypometabolism, ApoE genotype.

Method: Prospective multicentric study. 65 patients expected to enter the study.

Primary outcome measure: Standard Uptake Volume ratios.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Alzheimer's Disease (NINCDS-ADRDA) or from amnesic MCI
* 18 < MMS <= 28 for patients
* 28 <= MMS for healthy volunteers
* study period > 7 years
* native language : french
* signed informed consent
* affiliated to a social security system

Exclusion Criteria:

* alcoholism in medical history
* diabetes
* arterial hypertension (180/100 and more)
* chronical pulmonary disease with hypoxis
* cranial traumatism with loss of consciousness > 15 minutes
* severe depressive syndrome or anxiety
* psychiatric disease in medical history (excepted simple episodes of depression)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Standard Uptake Value Ratios (SUVr) | inclusion
  Standard Uptake Value Ratios (SUVr) in specific regions of interest (ROI) defined by the use of the cerebellum as reference region.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Camus, Principal Investigator — University Hospital of Tours
Locations (4):
- France (4):
  - university hospital of CAEN, Caen
  - University Hospital of Lille, Lille
  - University Hospital of Toulouse, Toulouse
  - University Hospital of Tours, Tours